CLINICAL TRIAL: NCT01080391
Title: A Randomized, Multicenter, Phase 3 Study Comparing Carfilzomib, Lenalidomide, and Dexamethasone (CRd) vs Lenalidomide and Dexamethasone (Rd) in Subjects With Relapsed Multiple Myeloma
Brief Title: Study Comparing Carfilzomib, Lenalidomide, and Dexamethasone (CRd) vs Lenalidomide and Dexamethasone (Rd) in Subjects With Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PX-171-009
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Results first posted 2015-07-08 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Relapsed Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Lenalidomide; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lenalidomide and Dexamethasone (Rd) (Active Comparator): Treatment was administered in cycles repeated every 28 days. Lenalidomide 25 mg was administered orally on days 1 to 21 and dexamethasone 40 mg was administered orally or IV on days 1, 8, 15, and 22.
  Interventions: Drug: Dexamethasone; Drug: Lenalidomide
- Carfilzomib, Lenalidomide, and Dexamethasone (CRd) (Experimental): Treatment was administered in cycles every 28 days. Carfilzomib 20 mg/m² was administered intravenously (IV) on days 1 and 2 of cycle 1, escalating to 27 mg/m² on days 8, 9, 15, and 16 of cycle 1 and continuing on days 1, 2, 8, 9, 15, and 16 of cycle 2 through cycle 12 and then from cycle 13 through cycle 18, 27 mg/m² on days 1, 2, 15, and 16. Lenalidomide 25 mg was administered orally on days 1 to 21 from cycle 1 through cycle 18 and from cycle 19 and higher. Dexamethasone 40 mg was administered orally or IV on days 1, 8, 15, and 22 from cycle 1 through cycle 18 and from cycle 19 and higher.
  Interventions: Drug: Dexamethasone; Drug: Lenalidomide; Drug: Carfilzomib

INTERVENTIONS:
Drug: Dexamethasone — 40 mg orally or IV on days 1, 8, 15, 22
Drug: Lenalidomide — 25 mg orally on days 1-21
  Other Names: Revlimid
Drug: Carfilzomib — 20 mg/m², 27 mg/m² intravenously
  Other Names: PR-171; Kyprolis®
  Arms: Carfilzomib, Lenalidomide, and Dexamethasone (CRd)

SUMMARY:
The primary objective was to compare progression-free survival in adults with relapsed multiple myeloma who are receiving CRd vs participants receiving Rd in a randomized multicenter setting.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, open-label, multicenter study comparing two treatment regimens for adults with relapsed multiple myeloma. Eligible subjects will be randomized in a 1:1 ratio to receive either the control Rd or CRd. Randomization will be stratified by β2 microglobulin levels (< vs ≥ 2.5 mg/L), prior bortezomib (no vs yes), and prior lenalidomide (no vs yes). Participants will receive the treatment determined by randomization in 28-day cycles until disease progression or unacceptable toxicity (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic multiple myeloma
2. Measurable disease, as defined by one or more of the following (assessed within 21 days prior to randomization):

   * Serum M-protein ≥ 0.5 g/dL
   * Urine Bence-Jones protein ≥ 200 mg/24 hours
   * For immunoglobulin A (IgA) patients whose disease can only be reliably measured by serum quantitative immunoglobulin (qIgA) ≥ 750 mg/dL (0.75 g/dL)
3. Prior treatment with at least one, but no more than three, regimens for multiple myeloma
4. Documented relapse or progressive disease on or after any regimen
5. Achieved a response to at least one prior regimen
6. Age ≥ 18 years
7. Life expectancy ≥ 3 months
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
9. Adequate hepatic function, with serum alanine aminotransferase (ALT) ≤ 3.5 times the upper limit of normal and serum direct bilirubin ≤ 2 mg/dL (34 µmol/L) within 21 days prior to randomization
10. Absolute neutrophil count ≥ 1.0 × 10^9/L within 21 days prior to randomization
11. Hemoglobin ≥ 8 g/dL (80 g/L) within 21 days prior to randomization
12. Platelet count ≥ 50 × 10^9/L (≥ 30 × 10^9/L if myeloma involvement in the bone marrow is > 50%) within 21 days prior to randomization
13. Creatinine clearance (CrCl) ≥ 50 mL/minute within 21 days prior to randomization
14. Written informed consent in accordance with federal, local, and institutional guidelines
15. Females of childbearing potential must agree to ongoing pregnancy testing and to practice contraception
16. Male subjects must agree to practice contraception

Exclusion Criteria:

1. If previously treated with bortezomib (alone or in combination), progression during treatment
2. If previously treated with a lenalidomide and dexamethasone (len/dex) combination:

   * Progression during the first 3 months of initiating treatment
   * Any progression during treatment if the len/dex combination was the subject's most recent line of therapy
3. Discontinuation of previous lenalidomide or dexamethasone due to intolerance; subjects intolerant to bortezomib are not excluded
4. Prior carfilzomib treatment
5. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
6. Waldenström's macroglobulinemia or IgM myeloma
7. Plasma cell leukemia (> 2.0 × 10^9/L circulating plasma cells by standard differential)
8. Chemotherapy or investigational agent within 3 weeks prior to randomization or antibody therapy within 6 weeks prior to randomization
9. Radiotherapy to multiple sites or immunotherapy/antibody therapy within 28 days prior to randomization; localized radiotherapy to a single site within 7 days prior to randomization
10. Corticosteroid therapy at a dose equivalent to dexamethasone > 4 mg/day within 21 days prior to randomization
11. Pregnant or lactating females
12. Major surgery within 21 days prior to randomization
13. Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to randomization
14. Known human immunodeficiency virus infection
15. Active hepatitis B or C infection
16. Myocardial infarction within 4 months prior to randomization, New York Hear Association (NYHA) Class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker
17. Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to randomization
18. Other malignancy, including myelodysplastic syndromes (MDS), within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
19. Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior to randomization
20. Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib)
21. Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment
22. Ongoing graft-vs-host disease
23. Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to randomization
24. Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 792 (Actual)
Dates: Start 2010-07-14 (Actual); Primary Completion 2014-06-16 (Actual); Study Completion 2017-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (127):
- United States (22):
  - Mayo Clinic, Scottsdale, Arizona
  - Providence St. Joseph Medical Center, Burbank, California
  - St. Jude Hospital Yorba Linda dba; St. Joseph Heritage Healthcare, Santa Rosa, California
  - Stanford University, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Cancer and Blood Disease Center, Lecanto, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Michigan - Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - NYU Clinical Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Associates in Oncology and Hematology, Chattanooga, Tennessee
  - The Don & Sybil Harrington Cancer Center, Amarillo, Texas
  - Baylor Sammons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin
- Austria (2):
  - Medizinische Universitat Wien, Vienna
  - Wilhelminspital der Stadt Wien, Zentrum fur Onkologie und Hamatologie, Vienna
- Belgium (6):
  - Ziekenhuisnetwerk Antwerpen - AZ Stuivenberg, Antwerp
  - AZ Sint-Jan AV, Bruges
  - Institut Jules Bordet, Brussels
  - UZ Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
- Bulgaria (5):
  - University Multiprofile Hospital for Active Treatment, "Dr. Georgi Stranski", Pleven
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi", Plovdiv
  - Military Medical Academy Multiprofile Hospital for Active Treatment, Sofia
  - Specialized Hospital for Active Treatment of Hematological Diseases, Sofia
  - Multiprofile Hospital for Active Treatment "Sveta Marina", Varna
- Canada (8):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - University of Alberta, Cross Cancer Institute, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - General Hospital, Health Sciences Centre, St. John's, Newfoundland and Labrador
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Health Center, Royal Victoria Hospital, Montreal, Quebec
  - Sir Mortimer B. Davis - Jewish General Hospital, Montreal, Quebec
- Czechia (5):
  - University Hospital Brno, Department of Internal Medicine - Hematooncology, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - University Hospital Kralovske Vinohrady - Prague, Prague
  - General University Hospital Prague, Prague
- France (9):
  - Hospital Antoine Beclere, Clamart
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans
  - Hopital Claude Huriez, Lille
  - CH de Mulhouse, Hopital Emile Muller, Mulhouse
  - CHU Nantes Hotel Dieu, Nantes
  - Hopital Saint-Antoine, Paris
  - Groupe Hospitalier Necker - Enfants Malades, Paris
  - Cancer Institut Universitaire de Toulouse-Oncopole (iUCT), Toulouse
  - Hopitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (8):
  - University of Dusseldorf, Düsseldorf
  - Krankenhaus Nordwest, Frankfurt am Main
  - University of Hamburg-Eppendorf, Hamburg
  - Universitat Heidelberg, Heidelberg
  - Stiftungsklinikum Mittelrhein, Koblenz
  - LMU Klinikum der Universitat, München
  - Universitatsklinikum Munster, Münster
  - Universitatsklinikum Wurzburg, Würzburg
- Greece (2):
  - Alexandra Hospital, Athens
  - University General Hospital of Patras, Pátrai
- Hungary (7):
  - St. Istvan and St. Laszlo Hospital of Budapest, Budapest
  - University of Debrecen, Medical and Health Science Center, Debrecen
  - Petz Aladar County Teaching Hospital, Győr
  - Bekes County Pandy Kalman Hospital, Gyula
  - Kaposi Mor County Teaching Hospital, Kaposvár
  - University of Pecs, Pécs
  - University of Szeged, Albert Szent-Gyorgi Clinical Center, Szeged
- Israel (6):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Ein Kerem, Jerusalem
  - Western Gailee Hospital - Nahariya, Nahariya
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
- Italy (5):
  - Azienda Ospedallera Niguarda Ca Granda, Milan
  - Azienda Ospedllero Maggiore della Carita, Novara
  - Azienda Ospedaliera Pisana Ospendale Santa Chiara - Main, Pisa
  - Ospedale S. Eugenio, Roma
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino
- Erasmus MC, Department of Haematology, Rotterdam, Netherlands
- Poland (8):
  - University Clinical Centre, Department of Hematologii Transplantologii, Gdansk
  - Samodzielny Publ. Szp. Wojewodzki w Gorzow Wlkp., Gorzów Wielkopolski
  - Independent Public Teaching Hospital of Medical University of Silesia in Katowice, Katowice
  - Nicolaus Copernicus Memorial Provincial Specialist Hospital in Lodz, Lodz
  - Szpital Wojewwodzki im. dr Ludwika Rydygiera w Suwalkach, Suwałki
  - Nicolaus Copernicus Municipal Specialist Hospital, Torun
  - Maria Sklodowska-Curie Institute of Oncology, Warsaw
  - Zamojski Non-Public Hospital, Zamość
- Romania (4):
  - Fundeni Clinical Institute, "Stefan Berceanu" Center for Hematology and Bone Marrow Transplantation, Bucharest
  - Coltea Clinical Hospital, Bucharest
  - Bucharest University Emergency Hospital, Bucharest
  - Regional Institute of Iasi, Iași
- Russia (9):
  - State Medical Institution Komi Republican Oncological Center, Syktyvkar, Komi
  - First Republican Clinical Hospital under the Ministry of Healthcare of the Republic of Udmurtia, Izhevsk
  - Federal State Budgetary Scientific Institution: N.N. Blokhin Russian Cancer Research Center, Moscow
  - Moscow State Medical Institution Municipal City Clinical Hospital n.a. S.P. Botkin, Moscow
  - Federal State Budget Institution: Hematology Research Center under MoH, Moscow
  - FSBI: Russian Research Institute of Hematology and Blood Transfusion under the Ferderal Agency for M&B, Saint Petersburg
  - State Higher Educational Institution: St Petersburg State Medical University n.a.I.P Pavlov, Saint Petersburg
  - SHEI: First St. Petersburg State Medical University N.a.I.P Pavlov under MoH, Clinic of Bone Marrow Transplant, Saint Petersburg
  - Federal State Budget Institute: Federal Almalov Medical Research Centre under Ministry of Healthcare, Saint Petersburg
- Serbia (5):
  - Clinical Center of Serbia, Clinic of Hematology, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Military Medical Academy, Clinic of Hematology, Belgrade
  - Clinical Center Nis, Clinic of Hematology, Niš
  - Clinical Center of Vojvodina, Clinic of Hematology, Novi Sad
- Spain (6):
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario y Politeecnico La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karolinska Universitetsjukhuset i Huddinge, Stockholm
  - Karolinska Universitetssjukhuset Solna, Hematologiskt Centrum, Stockholm
- United Kingdom (6):
  - St. Bartholomew's Hospital, London
  - Royal Free Hampstead, London
  - St. Georges Hospital, London
  - Nottingham University Hospitals (City Campus), Nottingham
  - Royal Marsden Hospital, Sutton
  - The Royal Wolverhampton Hospital NHS Trust, Wolverhampton

REFERENCES:
- [Background] Dimopoulos M, Wang M, Maisnar V, Minarik J, Bensinger W, Mateos MV, Obreja M, Blaedel J, Moreau P. Response and progression-free survival according to planned treatment duration in patients with relapsed multiple myeloma treated with carfilzomib, lenalidomide, and dexamethasone (KRd) versus lenalidomide and dexamethasone (Rd) in the phase III ASPIRE study. J Hematol Oncol. 2018 Apr 4;11(1):49. doi: 10.1186/s13045-018-0583-7. PMID 29615082
- [Background] Avet-Loiseau H, Fonseca R, Siegel D, Dimopoulos MA, Spicka I, Masszi T, Hajek R, Rosinol L, Goranova-Marinova V, Mihaylov G, Maisnar V, Mateos MV, Wang M, Niesvizky R, Oriol A, Jakubowiak A, Minarik J, Palumbo A, Bensinger W, Kukreti V, Ben-Yehuda D, Stewart AK, Obreja M, Moreau P. Carfilzomib significantly improves the progression-free survival of high-risk patients in multiple myeloma. Blood. 2016 Sep 1;128(9):1174-80. doi: 10.1182/blood-2016-03-707596. Epub 2016 Jul 20. PMID 27439911
- [Background] Dimopoulos MA, Stewart AK, Masszi T, Spicka I, Oriol A, Hajek R, Rosinol L, Siegel D, Mihaylov GG, Goranova-Marinova V, Rajnics P, Suvorov A, Niesvizky R, Jakubowiak A, San-Miguel J, Ludwig H, Ro S, Aggarwal S, Moreau P, Palumbo A. Carfilzomib-lenalidomide-dexamethasone vs lenalidomide-dexamethasone in relapsed multiple myeloma by previous treatment. Blood Cancer J. 2017 Apr 21;7(4):e554. doi: 10.1038/bcj.2017.31. PMID 28430175
- [Background] Dimopoulos MA, Stewart AK, Masszi T, Spicka I, Oriol A, Hajek R, Rosinol L, Siegel D, Mihaylov GG, Goranova-Marinova V, Rajnics P, Suvorov A, Niesvizky R, Jakubowiak A, San-Miguel J, Ludwig H, Palumbo A, Obreja M, Aggarwal S, Moreau P. Carfilzomib, lenalidomide, and dexamethasone in patients with relapsed multiple myeloma categorised by age: secondary analysis from the phase 3 ASPIRE study. Br J Haematol. 2017 May;177(3):404-413. doi: 10.1111/bjh.14549. Epub 2017 Feb 17. PMID 28211560
- [Background] Jakubowiak AJ, Campioni M, Benedict A, Houisse I, Tichy E, Giannopoulou A, Aggarwal SK, Barber BL, Panjabi S. Cost-effectiveness of adding carfilzomib to lenalidomide and dexamethasone in relapsed multiple myeloma from a US perspective. J Med Econ. 2016 Nov;19(11):1061-1074. doi: 10.1080/13696998.2016.1194278. Epub 2016 Jun 16. PMID 27224006
- [Background] Stewart AK, Dimopoulos MA, Masszi T, Spicka I, Oriol A, Hajek R, Rosinol L, Siegel DS, Niesvizky R, Jakubowiak AJ, San-Miguel JF, Ludwig H, Buchanan J, Cocks K, Yang X, Xing B, Zojwalla N, Tonda M, Moreau P, Palumbo A. Health-Related Quality-of-Life Results From the Open-Label, Randomized, Phase III ASPIRE Trial Evaluating Carfilzomib, Lenalidomide, and Dexamethasone Versus Lenalidomide and Dexamethasone in Patients With Relapsed Multiple Myeloma. J Clin Oncol. 2016 Nov 10;34(32):3921-3930. doi: 10.1200/JCO.2016.66.9648. PMID 27601539
- [Background] Chari A, Stewart AK, Russell SD, Moreau P, Herrmann J, Banchs J, Hajek R, Groarke J, Lyon AR, Batty GN, Ro S, Huang M, Iskander KS, Lenihan D. Analysis of carfilzomib cardiovascular safety profile across relapsed and/or refractory multiple myeloma clinical trials. Blood Adv. 2018 Jul 10;2(13):1633-1644. doi: 10.1182/bloodadvances.2017015545. PMID 29991494
- [Background] Facon T, Niesvizky R, Mateos MV, Siegel D, Rosenbaum C, Bringhen S, Weisel K, Ho PJ, Ludwig H, Kumar S, Wang K, Obreja M, Yang Z, Klippel Z, Mezzi K, Goldrick A, Tekle C, Dimopoulos MA. Efficacy and safety of carfilzomib-based regimens in frail patients with relapsed and/or refractory multiple myeloma. Blood Adv. 2020 Nov 10;4(21):5449-5459. doi: 10.1182/bloodadvances.2020001965. PMID 33166401
- [Background] Hari P, Mateos MV, Abonour R, Knop S, Bensinger W, Ludwig H, Song K, Hajek R, Moreau P, Siegel DS, Feng S, Obreja M, Aggarwal SK, Iskander K, Goldschmidt H. Efficacy and safety of carfilzomib regimens in multiple myeloma patients relapsing after autologous stem cell transplant: ASPIRE and ENDEAVOR outcomes. Leukemia. 2017 Dec;31(12):2630-2641. doi: 10.1038/leu.2017.122. Epub 2017 Apr 25. PMID 28439109
- [Background] Leleu X, Martin TG, Einsele H, Lyons RM, Durie BGM, Iskander KS, Ailawadhi S. Role of Proteasome Inhibitors in Relapsed and/or Refractory Multiple Myeloma. Clin Lymphoma Myeloma Leuk. 2019 Jan;19(1):9-22. doi: 10.1016/j.clml.2018.08.016. Epub 2018 Sep 5. PMID 30287200
- [Background] Mateos MV, Goldschmidt H, San-Miguel J, Mikhael J, DeCosta L, Zhou L, Obreja M, Blaedel J, Szabo Z, Leleu X. Carfilzomib in relapsed or refractory multiple myeloma patients with early or late relapse following prior therapy: A subgroup analysis of the randomized phase 3 ASPIRE and ENDEAVOR trials. Hematol Oncol. 2018 Apr;36(2):463-470. doi: 10.1002/hon.2499. Epub 2018 Feb 15. PMID 29446103
- [Background] Siegel DS, Dimopoulos MA, Ludwig H, Facon T, Goldschmidt H, Jakubowiak A, San-Miguel J, Obreja M, Blaedel J, Stewart AK. Improvement in Overall Survival With Carfilzomib, Lenalidomide, and Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma. J Clin Oncol. 2018 Mar 10;36(8):728-734. doi: 10.1200/JCO.2017.76.5032. Epub 2018 Jan 17. PMID 29341834
- [Background] Weisel K, Mateos MV, Gay F, Delforge M, Cook G, Szabo Z, Desgraz R, DeCosta L, Moreau P. Efficacy and safety profile of deep responders to carfilzomib-based therapy: a subgroup analysis from ASPIRE and ENDEAVOR. Leukemia. 2021 Jun;35(6):1732-1744. doi: 10.1038/s41375-020-01049-5. Epub 2020 Oct 16. PMID 33067574
- [Derived] Stewart AK, Rajkumar SV, Dimopoulos MA, Masszi T, Spicka I, Oriol A, Hajek R, Rosinol L, Siegel DS, Mihaylov GG, Goranova-Marinova V, Rajnics P, Suvorov A, Niesvizky R, Jakubowiak AJ, San-Miguel JF, Ludwig H, Wang M, Maisnar V, Minarik J, Bensinger WI, Mateos MV, Ben-Yehuda D, Kukreti V, Zojwalla N, Tonda ME, Yang X, Xing B, Moreau P, Palumbo A; ASPIRE Investigators. Carfilzomib, lenalidomide, and dexamethasone for relapsed multiple myeloma. N Engl J Med. 2015 Jan 8;372(2):142-52. doi: 10.1056/NEJMoa1411321. Epub 2014 Dec 6. PMID 25482145
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 14 July 2010 to 15 March 2012. The primary analysis was conducted using a data cut-off date of 16 June 2014 and the final safety analysis after last subject last visit date (05 December 2017).
Pre-assignment Details: Eligible participants were randomized in a 1:1 ratio to one of two treatment groups. Randomization was stratified by β2 microglobulin level (< vs. ≥ 2.5 mg/L), prior bortezomib exposure (no vs. yes), and prior lenalidomide exposure (no vs. yes).
Groups:
- Lenalidomide and Dexamethasone (Rd): Participants received their randomized study treatment in 28-day cycles until disease progression or unacceptable toxicity. Lenalidomide 25 mg was administered orally on days 1 to 21 and dexamethasone 40 mg was administered orally or intravenously on days 1, 8, 15, and 22.
- Carfilzomib, Lenalidomide, and Dexamethasone (CRd): Participants received their randomized study treatment in 28-day cycles until disease progression or unacceptable toxicity. Carfilzomib 20 mg/m² was administered intravenously (IV) on days 1 and 2 of cycle 1, then escalated to 27 mg/m² on Days 8, 9, 15, and 16 of cycle 1 and continuing on days 1, 2, 8, 9, 15, and 16 of cycle 2 through cycle 12 and then from cycle 13 through cycle 18, 27 mg/m² on days 1, 2, 15, and 16. Lenalidomide 25 mg was administered orally on days 1 to 21 of every cycle. Dexamethasone 40 mg was administered orally or IV on days 1, 8, 15, and 22 of every cycle.
Period: Overall Study
Arm/Group | Lenalidomide and Dexamethasone (Rd) | Carfilzomib, Lenalidomide, and Dexamethasone (CRd)
Started | 396 | 396
Treated | 389 | 392
Completed (Completed represents patients who discontinued treatment as of 05 December 2017) | 389 | 392
Not Completed | 7 | 4
Not completed — Randomized but not treated | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide and Dexamethasone (Rd) | Carfilzomib, Lenalidomide, and Dexamethasone (CRd) | Total
Number analyzed (Participants) | 396 | 396 | 792
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (9.04) | 63.3 (9.21) | 63.9 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 181 | 345
  Male | 232 | 215 | 447
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian/Native Hawaiian or Pacific Islander | 3 | 1 | 4
  Black or African American | 11 | 12 | 23
  White | 377 | 377 | 754
  Other | 4 | 6 | 10
Serum β2 Microglobulin [Count of Participants; unit: Participants]
  < 2.5 mg/L | 77 | 77 | 154
  ≥ 2.5 mg/L | 319 | 319 | 638
Prior Bortezomib Exposure [Count of Participants; unit: Participants]
  Yes | 261 | 261 | 522
  No | 135 | 135 | 270
Prior Lenalidomide Exposure [Count of Participants; unit: Participants]
  Yes | 78 | 80 | 158
  No | 318 | 316 | 634

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Kaplan-Meier estimate of median time from randomization to progressive disease (PD) or all-cause death. PD was assessed using International Myeloma Working Group-Uniform Response Criteria (IMWG-URC). One or more conditions were required to meet PD: 2 consecutive rising serum or urine M-protein from central lab; documented new bone lesion(s) or soft tissue plasmacytoma(s) or increased size of existing bone lesion(s) or plasmacytoma(s); or confirmed hypercalcemia due solely to plasma cell proliferative disorder (local lab greater than 11.5 mg/dL on 2 separate occasions). Censoring conditions (censoring dates) were: no post-baseline disease assessment (DA) (randomization date); started non-protocol systemic anticancer treatment before PD or death (last DA date before such treatment); died or had PD after more than 1 missed DA (last DA date without PD before the first missed visit); or were alive and without documentation of PD, including lost to follow-up without PD (last DA date).
Time Frame: From randomization through the data cutoff date of 16 June 2014. Median follow-up time was approximately 31 months.
Population: ITT analysis set comprised of all randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide and Dexamethasone (Rd) | Carfilzomib, Lenalidomide, and Dexamethasone (CRd)
Number analyzed (Participants) | 396 | 396
months | 17.6 [15.0 to 20.6] | 26.3 [23.3 to 30.5]
Statistical Analysis 1: Comparison: Lenalidomide and Dexamethasone (Rd) vs Carfilzomib, Lenalidomide, and Dexamethasone (CRd); Test type: Superiority or Other; p < 0.0001, Log Rank — Analysis was stratified by β2 microglobulin levels (< 2.5 mg/L vs. ≥ 2.5 mg/L), prior bortezomib (no vs. yes), and prior lenalidomide (no vs. yes); The stopping boundary for this analysis was 0.0127 based on 1-sided significance level (O'Brien-Fleming with Lan-DeMets spending function); Hazard Ratio (HR) = 0.690, 95% CI 2-sided [0.570 to 0.834]

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the duration from randomization to death due to any cause. Participants who were still alive were censored at the date when the participant was last known to be alive or the data cutoff date, whichever occurred earlier.
Time Frame: From randomization through the data cutoff date of 28 April 2017 for the final analysis of overall survival; median follow up time was 67.1 months in each treatment group.
Population: ITT analysis set comprised of all randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide and Dexamethasone (Rd) | Carfilzomib, Lenalidomide, and Dexamethasone (CRd)
Number analyzed (Participants) | 396 | 396
months | 40.4 [33.6 to 44.4] | 48.3 [42.4 to 52.8]
Statistical Analysis 1: Comparison: Lenalidomide and Dexamethasone (Rd) vs Carfilzomib, Lenalidomide, and Dexamethasone (CRd); The final analysis of OS was to be performed after 510 deaths occur. A total of 510 deaths would provide 85% power to detect, with a 1-sided significance level of 0.025, a hazard ratio of 0.765 corresponding to a 23.5% reduction in risk for death for CRd versus Rd (39.2 vs. 30.0 months, respectively); Test type: Superiority — The stopping boundary for this analysis was 0.0231 based on 1-sided significance level (O'Brien-Fleming with Lan-DeMets spending function); p = 0.0045, Log Rank; Analysis was stratified by β2 microglobulin levels (< 2.5 mg/L vs. ≥ 2.5 mg/L), prior bortezomib (no vs. yes), and prior lenalidomide (no vs. yes); Hazard Ratio (HR) = 0.794, 95% CI 2-sided [0.667 to 0.945]

3. Secondary Outcome: Overall Response Rate
Description: Overall response rate is defined as the percentage of participants who achieved either a confirmed stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) as their best response based on the Independent Review Committee (IRC) assessed response outcome. Response was determined using the International Myeloma Working Group - Uniform Response Criteria (IMWG-URC).
Time Frame: From randomization through the data cutoff date of 16 June 2014. Median follow-up time was approximately 31 months.
Population: ITT analysis set comprised of all randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide and Dexamethasone (Rd) | Carfilzomib, Lenalidomide, and Dexamethasone (CRd)
Number analyzed (Participants) | 396 | 396
percentage of participants | 66.7 [61.8 to 71.3] | 87.1 [83.4 to 90.3]
Statistical Analysis 1: Comparison: Lenalidomide and Dexamethasone (Rd) vs Carfilzomib, Lenalidomide, and Dexamethasone (CRd); Test type: Superiority; p < 0.0001, Cochran-Mantel Haenszel chi-square test; Cochran-Mantel Haenszel chi-square test with β2 macroglobulin level, prior bortezomib, and prior lenalidomide as stratification factors; Odds Ratio (OR) = 3.472, 95% CI 2-sided [2.411 to 5.001] — The odds ratio and 95% CI were estimated using the Mantel-Haenszel method

4. Secondary Outcome: Disease Control Rate
Description: Disease control rate was defined as the percentage of participants who achieved a best response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), minimal response (MR), or stable disease (SD) lasting ≥ 8 weeks according to International Myeloma Working Group - Uniform Response Criteria (IMWG-URC) (MR was determined using European Group for Blood and Marrow Transplantation criteria).
Time Frame: From randomization through the data cutoff date of 16 June 2014. Median follow-up time was approximately 31 months.
Population: ITT analysis set comprised of all randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide and Dexamethasone (Rd) | Carfilzomib, Lenalidomide, and Dexamethasone (CRd)
Number analyzed (Participants) | 396 | 396
percentage of participants | 87.1 [83.4 to 90.3] | 92.7 [89.7 to 95.0]
Statistical Analysis 1: Comparison: Lenalidomide and Dexamethasone (Rd) vs Carfilzomib, Lenalidomide, and Dexamethasone (CRd); Test type: Superiority; p = 0.0044, Cochran-Mantel Haenszel chi-square test; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.897, 95% CI 2-sided [1.17 to 3.08] — The odds ratio and 95% CI were estimated using the Mantel-Haenszel method

5. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) was calculated for participants who achieved a best response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR). Duration of response was defined as the time in months from the initial start of response (PR or better) to the earlier of documented progressive disease (PD) or death due to any cause. Participants who had not progressed or died were censored according to the censoring rules defined previously for PFS.
Time Frame: From randomization through the data cutoff date of 16 June 2014. Longest follow-up time was approximately 42 months.
Population: The Intent to treat (ITT) population with participantant who achieved a best overall response of PR or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide and Dexamethasone (Rd) | Carfilzomib, Lenalidomide, and Dexamethasone (CRd)
Number analyzed (Participants) | 264 | 345
months | 21.2 [16.7 to 25.8] | 28.6 [24.9 to 31.3]

6. Secondary Outcome: Duration of Disease Control
Description: Duration of disease control (DDC) was calculated for participants who achieved disease control. DDC was defined as the time in months from randomization to the earlier of documented progressive disease (PD) or death due to any cause. Participants who had not progressed or died were censored according to the censoring rules defined previously for PFS.
Time Frame: From randomization through the data cutoff date of 16 June 2014. Longest follow-up time was approximately 46 months.
Population: The Intent to treat (ITT) population with participantants who achieved disease control.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide and Dexamethasone (Rd) | Carfilzomib, Lenalidomide, and Dexamethasone (CRd)
Number analyzed (Participants) | 345 | 367
months | 18.9 [16.6 to 22.2] | 28.7 [24.4 to 31.6]

7. Secondary Outcome: Quality of Life Core Module (QLQ-C30) Global Health Status/Quality of Life Scores
Description: Health-related quality of life was assessed with the use of the European Organization for Research and Treatment of Cancer Quality of Life Core Module (QLQ-C30) questionnaire, a validated instrument in multiple myeloma patients. Scores range from 0 to 100, with higher scores indicating better health related quality of life.
Time Frame: Cycle 1 Day 1 (Baseline), Day 1 of Cycles 3, 6, 12, 18
Population: ITT analysis set participants with a baseline value.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lenalidomide and Dexamethasone (Rd) | Carfilzomib, Lenalidomide, and Dexamethasone (CRd)
Number analyzed (Participants) | 367 | 375
scores on a scale
  Cycle 1 Day 1 (Baseline) | 58.1 (21.7) | 58.3 (21.7)
  Cycle 3, Day 1: number analyzed (Participants) | 334 | 356
  Cycle 3, Day 1 | 56.8 (19.4) | 59.9 (20.4)
  Cycle 6, Day 1: number analyzed (Participants) | 284 | 326
  Cycle 6, Day 1 | 58.9 (19.7) | 62.5 (20.1)
  Cycle 12, Day 1: number analyzed (Participants) | 212 | 255
  Cycle 12, Day 1 | 57.3 (19.7) | 62.7 (19.6)
  Cycle 18, Day 1: number analyzed (Participants) | 147 | 226
  Cycle 18, Day 1 | 59.9 (18.8) | 64.3 (19.2)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug to 30 days after the last dose or initiation of new anticancer therapy, whichever occurred first. Median treatment duration was 57 and 88 weeks in each treatment group respectively, with a maximum of 338 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Lenalidomide and Dexamethasone (Rd) | Carfilzomib, Lenalidomide, and Dexamethasone (CRd)
Serious Adverse Events (participants affected / at risk) | 221/389 | 256/392
Other Adverse Events (participants affected / at risk) | 358/389 | 370/392
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide and Dexamethasone (Rd) (N=389) | Carfilzomib, Lenalidomide, and Dexamethasone (CRd) (N=392)
Anaemia (Blood and lymphatic system disorders) | 10 | 8
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 8
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 5 | 4
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Platelet disorder (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 5
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 5
Angina pectoris (Cardiac disorders) | 4 | 2
Angina unstable (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 8 | 9
Atrial flutter (Cardiac disorders) | 1 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 3 | 5
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 3 | 5
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 2
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 2
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 6
Myocardial ischaemia (Cardiac disorders) | 0 | 2
Pericardial effusion (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 5
Cataract nuclear (Eye disorders) | 1 | 0
Cataract subcapsular (Eye disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 7
Diverticular perforation (Gastrointestinal disorders) | 0 | 2
Diverticulum oesophageal (Gastrointestinal disorders) | 0 | 1
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 0 | 2
Chest pain (General disorders) | 1 | 1
Death (General disorders) | 2 | 2
Disease progression (General disorders) | 8 | 4
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 4 | 0
Influenza like illness (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 9 | 14
Sudden death (General disorders) | 1 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 3 | 4
Cholelithiasis (Hepatobiliary disorders) | 1 | 2
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 2
Bacterial infection (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 11 | 9
Bronchitis viral (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 7 | 5
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 4 | 1
Cholangitis suppurative (Infections and infestations) | 0 | 1
Chronic hepatitis C (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 4
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 3
Diverticulitis (Infections and infestations) | 1 | 1
Endocarditis (Infections and infestations) | 0 | 2
Enterocolitis bacterial (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 5 | 5
Genitourinary tract infection (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 0 | 1
Hepatic infection (Infections and infestations) | 1 | 0
Herpes zoster disseminated (Infections and infestations) | 1 | 1
Incision site infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 2 | 3
Laryngitis bacterial (Infections and infestations) | 0 | 1
Listeria sepsis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 3 | 2
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 3
Neutropenic sepsis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 52 | 67
Pneumonia bacterial (Infections and infestations) | 3 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 8 | 16
Respiratory tract infection viral (Infections and infestations) | 2 | 1
Salmonella sepsis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 5 | 7
Sepsis syndrome (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 4 | 3
Sinusitis (Infections and infestations) | 2 | 4
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 1
Testicular abscess (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 2
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 2 | 4
Urosepsis (Infections and infestations) | 2 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 3 | 5
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 2
Gallbladder injury (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 3 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Splenic injury (Injury, poisoning and procedural complications) | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1
Cardiac stress test abnormal (Investigations) | 0 | 1
General physical condition abnormal (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Influenza A virus test positive (Investigations) | 0 | 2
Intraocular pressure increased (Investigations) | 0 | 1
Monoclonal immunoglobulin present (Investigations) | 0 | 1
Respiratory syncytial virus test positive (Investigations) | 0 | 1
Streptococcus test positive (Investigations) | 0 | 1
Viral test positive (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Mineral deficiency (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 3
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemia plasmacytic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Altered state of consciousness (Nervous system disorders) | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 1
Cerebral cyst (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 10 | 4
Cognitive disorder (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 2 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Hydrocephalus (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Myxoedema coma (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 3 | 2
Syncope (Nervous system disorders) | 2 | 3
Transient ischaemic attack (Nervous system disorders) | 3 | 0
VIth nerve paralysis (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Disorientation (Psychiatric disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 1 | 0
Personality change (Psychiatric disorders) | 0 | 1
Psychiatric decompensation (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 4 | 6
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 12
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 4
Aortic aneurysm (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 6 | 9
Embolism (Vascular disorders) | 0 | 2
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 3
Vasculitis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Cardiac asthma (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Disease progression (General disorders) | 8 | 5
Drowning (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 4 | 2
Multiple organ dysfunction syndrome (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 3
Pyrexia (General disorders) | 12 | 15
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1
Cholangitis infective (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 2
Epididymitis (Infections and infestations) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Osteomyelitis bacterial (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Stoma site abscess (Infections and infestations) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 8
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Urethral prolapse (Renal and urinary disorders) | 0 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide and Dexamethasone (Rd) (N=389) | Carfilzomib, Lenalidomide, and Dexamethasone (CRd) (N=392)
Anaemia (Blood and lymphatic system disorders) | 154 | 166
Leukopenia (Blood and lymphatic system disorders) | 22 | 33
Neutropenia (Blood and lymphatic system disorders) | 133 | 157
Thrombocytopenia (Blood and lymphatic system disorders) | 94 | 115
Cataract (Eye disorders) | 36 | 39
Vision blurred (Eye disorders) | 15 | 24
Abdominal pain (Gastrointestinal disorders) | 27 | 32
Abdominal pain upper (Gastrointestinal disorders) | 12 | 28
Constipation (Gastrointestinal disorders) | 69 | 81
Diarrhoea (Gastrointestinal disorders) | 143 | 170
Dyspepsia (Gastrointestinal disorders) | 22 | 24
Nausea (Gastrointestinal disorders) | 57 | 82
Vomiting (Gastrointestinal disorders) | 34 | 49
Asthenia (General disorders) | 56 | 69
Chills (General disorders) | 9 | 25
Fatigue (General disorders) | 119 | 128
Oedema peripheral (General disorders) | 75 | 85
Pyrexia (General disorders) | 78 | 105
Bronchitis (Infections and infestations) | 56 | 75
Influenza (Infections and infestations) | 14 | 26
Nasopharyngitis (Infections and infestations) | 65 | 87
Pneumonia (Infections and infestations) | 29 | 45
Respiratory tract infection (Infections and infestations) | 39 | 41
Sinusitis (Infections and infestations) | 18 | 24
Upper respiratory tract infection (Infections and infestations) | 81 | 115
Urinary tract infection (Infections and infestations) | 21 | 36
Viral infection (Infections and infestations) | 11 | 28
Alanine aminotransferase increased (Investigations) | 15 | 21
Blood creatinine increased (Investigations) | 21 | 27
Neutrophil count decreased (Investigations) | 22 | 21
Decreased appetite (Metabolism and nutrition disorders) | 35 | 47
Hyperglycaemia (Metabolism and nutrition disorders) | 39 | 48
Hypocalcaemia (Metabolism and nutrition disorders) | 49 | 65
Hypokalaemia (Metabolism and nutrition disorders) | 58 | 114
Hypomagnesaemia (Metabolism and nutrition disorders) | 29 | 40
Hypophosphataemia (Metabolism and nutrition disorders) | 33 | 57
Arthralgia (Musculoskeletal and connective tissue disorders) | 57 | 57
Back pain (Musculoskeletal and connective tissue disorders) | 81 | 73
Bone pain (Musculoskeletal and connective tissue disorders) | 36 | 39
Muscle spasms (Musculoskeletal and connective tissue disorders) | 82 | 106
Muscular weakness (Musculoskeletal and connective tissue disorders) | 24 | 28
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 29 | 26
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 36 | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 22 | 25
Pain in extremity (Musculoskeletal and connective tissue disorders) | 42 | 48
Dizziness (Nervous system disorders) | 45 | 54
Dysgeusia (Nervous system disorders) | 21 | 14
Headache (Nervous system disorders) | 32 | 56
Neuropathy peripheral (Nervous system disorders) | 28 | 34
Paraesthesia (Nervous system disorders) | 23 | 27
Peripheral sensory neuropathy (Nervous system disorders) | 27 | 25
Tremor (Nervous system disorders) | 32 | 28
Anxiety (Psychiatric disorders) | 17 | 33
Insomnia (Psychiatric disorders) | 65 | 81
Cough (Respiratory, thoracic and mediastinal disorders) | 70 | 116
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 59 | 76
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 19 | 23
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 | 28
Erythema (Skin and subcutaneous tissue disorders) | 13 | 30
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 18 | 28
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 31
Rash (Skin and subcutaneous tissue disorders) | 59 | 50
Deep vein thrombosis (Vascular disorders) | 11 | 21
Hypertension (Vascular disorders) | 30 | 62
Hypotension (Vascular disorders) | 22 | 26
Toothache (Gastrointestinal disorders) | 12 | 20
Asthenia (General disorders) | 57 | 72
Chills (General disorders) | 9 | 26
Fatigue (General disorders) | 124 | 132
Oedema peripheral (General disorders) | 66 | 78
Peripheral swelling (General disorders) | 21 | 21
Pyrexia (General disorders) | 80 | 110
Viral upper respiratory tract infection (Infections and infestations) | 68 | 80
Weight decreased (Investigations) | 20 | 14
Hyperuricaemia (Metabolism and nutrition disorders) | 11 | 22
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 | 20
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.